CLINICAL TRIAL: NCT06697002
Title: Effects of Lower Trapezius Strengthening Versus Scapular Mobility Exercise on Pain, Range of Motion and Disability Among Snooker Players in Unilateral Neck Pain
Brief Title: Effects of Lower Trapezius Strengthening Versus Scapular Mobility Exercise Among Snooker Players in Unilateral Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0405
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: Disability; Lower trapezius strength; Strengthening exercise; Mobility exercise; unilateral neck pain

STUDY DESIGN:
Intervention Model Description: randomized control design
Who Masked: Participant
Masking Description: the participants are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 32 participants will be in control group,they will only perform lower tapezius strenghtening excercise and will not perform scapular mobility excercises.
  Interventions: Other: lower trapezius strenghtening excercise
- Group B (Experimental): 32 participants will be in experimental group,they will perform scapular mobility excercise
  Interventions: Other: scapular mobility exercise

INTERVENTIONS:
Other: lower trapezius strenghtening excercise — 32 participants will be in control group who will perform strenghtening excerise of lower trapezius
  Arms: Group A
Other: scapular mobility exercise — 32 participants will be in experimental group who will perform scapular mobility exercise
  Arms: Group B

SUMMARY:
Effects of lower trapezius strengthening versus scapular mobility exercise among snooker players in unilateral neck pain.

DETAILED DESCRIPTION:
Effects of lower trapezius strengthening versus scapular mobility exercise on pain, range of motion and disability among snooker players in unilateral neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 35 years,
* Males snooker players
* Neck pain perceived by individual as being on one side of the neck Pain 3 or more month in duration.
* Participants with 6-7 level of pain on NPRS scale
* Participants with scapular mobility limited

Exclusion Criteria:

* Neck pain perceived by individual as being centrally located or on both sides of neck.
* Radicular symptoms
* History of cervical spine surgery
* Traumatic neck injury
* underlying neurological condition

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
NECK DISABILITY INDEX (NDI SCALE) | 8 weeks
  Each section of NDI is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.
  Points summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability. it should be noted before exercise and after 8 week of exercise in uni lateral neck pain players .
  BENCHMARK FOUND; 1.0-4points (0-8%) no disability, 2.5-14points ( 10 - 28%) mild disability, 3.15-24points (30-48% ) moderate disability, 4.25-34points (50- 64%) severe disability, 5.35-50points (70-100%) complete disability
NPRS | 8 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a uni-dimensional measure of pain intensity in adults with chronic pain.
  the 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  we measure snooker players pain on a scale before exercise and after exercise to find pretest and posttest pain intensity.
GONIOMETER | 8 weeks
  we measure cervical range of motion in flexion and extension through goniometer before performing exercise and after strenghtening and mobility exercise

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoor samad, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- LDA sports complex, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sjogaard G, Sogaard K, Hansen AF, Ostergaard AS, Teljigovic S, Dalager T. Exercise Prescription for the Work-Life Population and Beyond. J Funct Morphol Kinesiol. 2023 May 26;8(2):73. doi: 10.3390/jfmk8020073. PMID 37367237
- [Background] Ahmed H, Jarrar MA, Ahmed R, Alqhtani R, Alshahrani A. Effect of Post-Isometric Relaxation and Laser on Upper Trapezius Trigger Point Pain in Patients with Mechanical Neck Pain. Niger J Clin Pract. 2020 Dec;23(12):1660-1666. doi: 10.4103/njcp.njcp_6_20. PMID 33355818
- [Background] Alghadir AH, Iqbal A, Anwer S, Iqbal ZA, Ahmed H. Efficacy of Combination Therapies on Neck Pain and Muscle Tenderness in Male Patients with Upper Trapezius Active Myofascial Trigger Points. Biomed Res Int. 2020 Mar 10;2020:9361405. doi: 10.1155/2020/9361405. eCollection 2020. PMID 32258159
- [Background] Wang DM, Li C, Hatchard N, Chang Chien GC, Alm J. Lower trapezius muscle function in people with and without shoulder and neck pain: a systematic review. J Osteopath Med. 2022 Sep 13;123(2):73-89. doi: 10.1515/jom-2022-0056. eCollection 2023 Jan 1. PMID 36100364
- [Background] Grassini S. Virtual Reality Assisted Non-Pharmacological Treatments in Chronic Pain Management: A Systematic Review and Quantitative Meta-Analysis. Int J Environ Res Public Health. 2022 Mar 29;19(7):4071. doi: 10.3390/ijerph19074071. PMID 35409751
- [Background] Javdaneh N, Saeterbakken AH, Shams A, Barati AH. Pain Neuroscience Education Combined with Therapeutic Exercises Provides Added Benefit in the Treatment of Chronic Neck Pain. Int J Environ Res Public Health. 2021 Aug 22;18(16):8848. doi: 10.3390/ijerph18168848. PMID 34444594
- [Background] van de Wijdeven B, Visser B, Kuijer PPFM. Evaluating the categorisation of interventions in individual working practice aimed at preventing work-related musculoskeletal disorders: An international experts consultation. Appl Ergon. 2024 Oct;120:104338. doi: 10.1016/j.apergo.2024.104338. Epub 2024 Jul 4. PMID 38968738
- [Background] Pan JW, Mei Q, Fernandez J, Song H, Komar J, Kong PW. Computer simulation on the cueing movements in cue sports: a validation study. PeerJ. 2023 Oct 11;11:e16180. doi: 10.7717/peerj.16180. eCollection 2023. PMID 37842036
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399